CLINICAL TRIAL: NCT01566916
Title: Medium Term Survivorship of Cementless THA Performed Using the Bone Preservation Tri-Lock Femoral Stem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RIFJPAR 12-01
Record Dates: First submitted 2012-02-24; First posted 2012-03-29 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

ARMS (2):
- Total Hip Arthroplasty performed via direct anterior approach (Active Comparator)
  Interventions: Procedure: Total Hip Arthroplasty
- Total Hip Arthroplasty using anterolateral approach (Active Comparator)
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty

SUMMARY:
This prospective, randomized study will study the 2 year survivorship and short term outcomes of a currently-used femoral stem: the Bone Preservation Tri-Lock femoral stem using two surgical approaches. The surgical approaches being studied are direct anterior and anterolateral. Implant survivorship, radiographic positioning, and functional outcomes will be compared. Subjects will be randomized to surgical approach and followed for a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed an IRB, study specific informed patient consent
* Patient is a male or non-pregnant female age 21 years or older at the time of study device implantation
* Patient has primary diagnosis of non-inflammatory degenerative joint disease.
* Patient is a candidate for primary cementless total hip replacement
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) > 40 Kg/m2
* Patient has an active or suspected infection at the time of device implantation
* Patient is immunologically suppressed.
* Patient requires revision surgery of a previously implanted total hip replacement
* Patient has a known sensitivity to device materials

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Survivorship of Bone Preservation Tri-Lock femoral stem | 2 years post-op
  Survivorship will be assessed via radiographic (x-ray) analysis and need for revision surgery (if patient had femoral stem removed for any reason within the first two years after surgery).

SECONDARY OUTCOMES:
TUG (timed up and go) Score | 6 weeks post-op

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rothman Institute, Egg Harbor, New Jersey
  - Rothman Institute, Philadelphia, Pennsylvania